CLINICAL TRIAL: NCT06636630
Title: Evaluating the Efficacy of Double Flap Versus Quadruple Flap Techniques in Stabilizing Ball Implants Post-Evisceration: a Comparative Analysis
Brief Title: Comparing Double VS Quadruple Flap for Securing Ball Implants After Eye Ball Evisceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Khaled Kotb Abdallah, Lecturer of ophthalmology fayoum university, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fayoum university hospital
Record Dates: First submitted 2024-10-09; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Evisceration; Traumatic, Eye
Keywords: Evisceration, Ball implants, Double flap technique, Quadruple flap technique.

STUDY DESIGN:
Intervention Model Description: The study will enroll patients requiring evisceration with implant placement due to conditions such as end-stage painful blind eye, intraocular tumors, or severe ocular trauma. Patients will be randomly assigned to one of two surgical techniques: Double Flap Technique (Group A) or Quadriple Flap Technique (Group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double scleral flap (Experimental): Double Flap Technique (Group A) A 360-degree peritomy will be performed to expose the underlying sclera. Following evisceration of the ocular contents, careful hemostasis will be achieved. Two muscular-tendinous flaps will be developed from the horizontal rectus muscles. These flaps will be dissected under minimal tension to preserve their vascular supply. The prepared flaps will be draped over the implant in a manner that the edges slightly overlap, ensuring complete coverage. The flaps will be sutured together using silk sutures, securing the implant in place.The conjunctiva will be meticulously closed over the muscle flaps with continuous absorbable sutures to enhance the healing process and minimize postoperative discomfort.
  Interventions: Procedure: Double scleral flap
- Quadruple scleral flap (Experimental): Quadruple flap technique involves creating four scleral flaps, which proponents argue provides a more robust framework for securing the implant. This technique is designed to enhance the integration of the implant with surrounding orbital structures, thereby potentially reducing the risk of exposure and improving cosmetic outcomes. The quadruple flap method is suggested to better preserve the orbital anatomy, allowing for superior distribution of volume and more natural prosthetic motility.
  Interventions: Procedure: Quadruple scleral flap

INTERVENTIONS:
Procedure: Quadruple scleral flap — Quadruple Flap Technique (Group B) A 360-degree peritomy will be performed to expose the underlying sclera. Following evisceration of the ocular contents, careful hemostasis will be achieved. Four muscular-tendinous flaps will be developed from the recti muscles. These flaps will be dissected under minimal tension to preserve their vascular supply. The prepared flaps will be draped over the implant in a manner that the edges slightly overlap, ensuring complete coverage. The flaps will be sutured together using silk sutures, securing the implant in place.The conjunctiva will be meticulously closed over the muscle flaps with continuous absorbable sutures to enhance the healing process and minimize postoperative discomfort.
  Arms: Quadruple scleral flap
Procedure: Double scleral flap — The double flap technique, which involves the creation of two scleral flaps to encase and secure the implant, has been a standard approach in many surgical settings. This method aims to cover the implant adequately, thereby minimizing exposure risks and enhancing the potential for implant motility.
  Arms: Double scleral flap

SUMMARY:
The primary objective of this interventional study is to compare the efficacy and outcomes of the double flap and quadruple flap closure techniques in securing ball implants after evisceration. Specific objectives include:

1. Assessing the rate of implant migration and extrusion.
2. Evaluating the long-term stability of the implant within the scleral shell.
3. Investigating the occurrence of complications such as exposure or infection.
4. Analyzing the functional and anatomical outcomes of the closure techniques.
5. Comparing patient satisfaction and quality of life measures.

DETAILED DESCRIPTION:
The choice of surgical technique for stabilizing ball implants following evisceration has a significant impact on both functional and aesthetic outcomes for patients. Evisceration, a procedure that involves the removal of intraocular contents while preserving the scleral shell and extraocular muscles, is typically performed to alleviate pain in a blind eye, prevent sympathetic ophthalmia, or improve the cosmetic appearance of a disfigured eye (Shields et al. 2022). Ball implants are commonly used to restore the anatomic integrity and appearance of the orbit post-evisceration, but their success largely depends on the stability provided by the surgical technique employed (Wang et al. 2023).

Recent advancements in oculoplastic surgery have introduced several techniques to enhance implant stability, with the double flap and quadruple flap methods gaining particular attention. The double flap technique involves the use of two scleral flaps to secure the implant, while the quadruple flap method utilizes four flaps to provide greater coverage and stability (Singh et al. 2023). Despite the increasing popularity of these techniques, there remains a lack of consensus regarding their relative efficacy in ensuring implant stability and minimizing complications, such as migration, exposure, or extrusion of the implant (Patel et al. 2023).

Some studies suggest that the quadruple flap technique offers superior stability due to increased tissue coverage, potentially reducing the risk of postoperative complications (Gonzalez et al. 2024). However, other research indicates that the double flap technique is equally effective, with the added benefit of reduced operative time and fewer intraoperative adjustments (Harrison et al. 2023). Given these conflicting findings, there is a clear need for further investigation to determine the most effective approach for stabilizing ball implants post-evisceration.

This study aims to evaluate and compare the efficacy of the double flap and quadruple flap techniques in stabilizing ball implants following evisceration.

Patients and Methods This prospective, randomized, controlled trial was conducted at the Department of Ophthalmic Surgery, Faculty of Medicine, Fayoum University during the period from January 2024 to July 2024. Approval was granted by the institutional ethics committee, adhered to the tenets of the Declaration of Helsinki and informed consent was secured from all participants.

Participants included patients requiring evisceration with implant placement due to conditions such as end-stage painful blind eye and endophthalmitis. All participants were randomly assigned to undergo either the Quadruple Flap Technique (Group A) or the Double Flap Technique (Group B). Eligible participants were 18 years or older, diagnosed with conditions necessitating evisceration with implant placement, and able to provide informed consent. Patients with previous ocular surgeries affecting orbital anatomy, systemic conditions influencing wound healing, or allergies to implant materials were excluded from the study.

Initial Assessment and Diagnostic Testing All patients underwent an initial consultation, which included a comprehensive medical and ocular history to identify any risk factors that could impact the surgery or the choice of implant, such as prior ocular procedures, systemic diseases, or allergies. A thorough physical examination was conducted, with a focus on the ocular area to assess the condition of the eye and surrounding tissues. Ultrasound was used to assess the integrity of the ocular structures, plan implant size and confirm the diagnosis.

Ophthalmic Assessment and Patient Counseling Each patient received a comprehensive ophthalmic assessment, which involved documentation of any remaining visual function, examination of the eyelids, conjunctiva, and cornea, and measurement of intraocular pressure to evaluate overall eye health. Silicone implant was used for all patients, and the appropriate size and shape of the implant were determined based on the patient's orbital volume and anatomy. Counseling sessions were conducted to provide detailed information about the selected surgical procedure, its risks and benefits, and postoperative expectations. Written informed consent was obtained from all participants after ensuring they fully understood the procedure and had the opportunity to ask questions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with conditions necessitating evisceration with implant
* Able to provide informed consent

Exclusion Criteria:

* Previous ocular surgery affecting orbital anatomy
* Systemic conditions influencing wound healing (e.g., diabetes, autoimmune disorders)
* Allergy to implant materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluating the post-operative extrusion rates of the ball implant from the scleral shell | Through study completion, an average of 6 months
  The primary outcome measure was implant stability, assessed clinically and through imaging at 1, 3, and 6 months postoperatively to review any signs of implant migration or extrusion as well as signs of conjunctival erosion.

SECONDARY OUTCOMES:
Postoperative pain | From enrollment to the end of the follow up period after 6 months
  The Quality of Life (VAS) Score was determined using a Visual Analog Scale,
Postoperative complications | From enrollment to the end of the follow up period after 6 months
Patient satisfaction with implant motility | From enrollment to the end of the follow up period after 6 months
  Assessed through a standardized questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum university hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No